CLINICAL TRIAL: NCT04670952
Title: The Pulmonary Effects of Low Pressure Versus Standard Pressure Laparoscopic Cholecystectomy in Patients With Cardiopulmonary Disorders: A Prospective Randomized Controlled Trial
Brief Title: Potential Pulmonary Benefit of Low Pressure Laparoscopic Cholecystectomy in Selected Patients
Acronym: POPLOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Feng Tian, Attending, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Feng Tian
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Cholecystitis/Cholelithiasis; Cholecystitis; Gallstone; Polyp Gallbladder
Keywords: low pressure; laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis; Cholelithiasis; Gallstones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: It will be single blinded. Operator, first assistant and data collector could not be blinded. Whereas patients, nurses, data analyzer, and those who have the access to the primary predictor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Pressure Laparoscopic Cholecystectomy (Experimental): LPLC refers to "Low Pressure Laparoscopic Cholecystectomy". In this arm, the pneumoperitoneum pressure is set as 10mmHg.
  Interventions: Other: Low Pressure Laparoscopic Cholecystectomy
- Standard Pressure Laparoscopic Cholecystectomy (Other): This is taken as the control group. SPLC refers to "Standard Pressure Laparoscopic Cholecystectomy". In this arm, the pneumoperitoneum pressure is set as 14 mmHg.
  Interventions: Other: Standard Pressure Laparoscopic Cholecystectomy

INTERVENTIONS:
Other: Low Pressure Laparoscopic Cholecystectomy — Low Pressure Laparoscopic Cholecystectomy (10mmHg) is set as the experimental group.
  Arms: Low Pressure Laparoscopic Cholecystectomy
Other: Standard Pressure Laparoscopic Cholecystectomy — Standard Pressure Laparoscopic Cholecystectomy (14mmHg) is set as the control group.
  Arms: Standard Pressure Laparoscopic Cholecystectomy

SUMMARY:
Standard Pressure Laparoscopic Cholecystectomy，as the standard for cholecystectomy, can lead to about 15% of pulmonary atelectasis. According to literature, low pressure laparoscopic cholecystectomy is thought to probably decrease cardio-pulmonary related complications and postoperative pain. However, the previous studies have presented controversial results. Our study aim to evaluate the potential pulmonary benefit of low pressure laparoscopic cholecystectomy in elderly or patients accompanied with cardio-pulmonary disorders.

DETAILED DESCRIPTION:
Standard Pressure Laparoscopic Cholecystectomy, SPLC；12-16mmHg，as the standard for cholecystectomy, can lead to about 15% of pulmonary atelectasis.

According to literature, Low Pressure Laparoscopic Cholecystectomy, LPLC；8-10mmHg is thought to probably decrease cardio-pulmonary related complications and postoperative pain. However, most of the existing study have combined population with all age scale, bringing bias to the result. Our study aim to evaluate the potential pulmonary benefit of low pressure laparoscopic cholecystectomy in elderly or patients accompanied with cardio-pulmonary disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85;
2. Patients receiving laparoscopic cholecystectomy due to benign gallbladder diseases;
3. Older patient or accompanied by cardiopulmonary diseases (age>60 years, hypertension, Diabetes Mellitus, coronary heart disease, arrhythmia, chronic bronchitis, emphysema, history of heart surgery, history of lung surgery, history of mediastinal surgery, asthma, et al);
4. Aged older than 60, with or without the above diseases;
5. American society of Aneshesiologists (ASA) II or higher;
6. Informed consent acquired.

Exclusion Criteria:

1. Having contraindication of laparoscopic operations;
2. History at epigastric surgery. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of partial pressure of carbon dioxide（pCO2） | Within postoperative 30 days.
  Change of pCO2 in arterial blood gas test

SECONDARY OUTCOMES:
operation time | During surgery.
  skin to skin operative duration
conversion rate to open surgery | During surgery.
  Need of conversion to open surgery duo to adhesion, hemorrhage, or other reasons.
visual analogue scale (VAS) | During postoperative 24 hours.
  For evaluation of postoperative pain degree, using VAS, scoring 1-10 scores.
complication rate | Within postoperative 30 days.
  Rate of total postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong He, Doctor, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian F, Sun X, Yu Y, Zhang N, Hong T, Liang L, Yao B, Song L, Pei C, Wang Y, Lu W, Qu Q, Guo J, Zhang T, He X. Comparison of low-pressure and standard-pressure pneumoperitoneum laparoscopic cholecystectomy in patients with cardiopulmonary comorbidities: a double blinded randomized clinical trial. BMC Surg. 2024 Nov 6;24(1):348. doi: 10.1186/s12893-024-02606-w. PMID 39506748